CLINICAL TRIAL: NCT03750318
Title: Validation Study on RENEW's Aingeal at KK Women's and Children's Hospital
Acronym: RENEW
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Renew Group (Industry)
Responsible Party: Principal Investigator, Sng Ban Leong, Head and Senior Consultant, Dept of Women's Anaesthesia, KK Women's and Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018/2223 (Women)
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Vital Sign; Heart Rate; Respiratory Rate
Keywords: Vital sign monitoring; Heart rate; Respiratory rate

STUDY DESIGN:
Intervention Model Description: All patients recruited will be wearing the Aingeal device as part of an integrated monitoring with opioid delivery system at ward setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Aingeal (Experimental): All patients will wear the Aingeal device as part of the vital sign monitoring with opioid delivery system at ward setting.
  Interventions: Device: Vital sign monitoring

INTERVENTIONS:
Device: Vital sign monitoring — Each patient will be set up for monitoring on admission. Duration of opioid therapy for post-operative in-patients may range from 1-3 days. Once opioid therapy is no longer required, Aingeal monitoring will be ended and each patient would be encouraged to have at least 1 day Aingeal monitoring to be recorded during the study. De-identified log files will be extracted from the Surveillance Station and reprocessed to produce counts of the number of alarms raised during monitoring. A sample of the data will be reviewed to determine whether cardiac and respiratory alarms are defined as True or False, with an overall Alarm Rate per patient per day and False Positive Alarm Rate per patient per day derived. Vital sign trend graphs for each patient will be produced.

SUMMARY:
This proposal describes the evaluation of a CE-marked, FDA cleared vital signs Surveillance Monitoring system within an adult in-patient setting KK Women's and Children's Hospital ("KKH"), the main tertiary women and children hospital in Singapore. User acceptance of Aingeal and the Surveillance System will be considered within the clinical settings.

DETAILED DESCRIPTION:
RENEW's Surveillance Monitoring system is made up of two main components: a patient-worn wireless vital signs monitor (Aingeal) that transmits data over Wi-Fi to a central station software platform (Surveillance Station). The Aingeal device measures single lead ECG, heart rate, respiration waveform and rate, and skin temperature. A snapshot of data is transmitted by the devices intermittently to the Surveillance Station, enabling vital signs trends to be plotted. If any heart, respiration rate or skin temperature values move outside of pre-defined high and low limits (individually set for each patient) an alert is raised. ECG arrhythmia detection algorithms automatically record and send ECG data if the patient is suspected to be experiencing an arrhythmia event (Asystole, Ventricular Fibrillation, Tachycardia or Bradycardia). This proposal describes the evaluation of RENEW's Aingeal device within an adult in-patient setting KK Women's and Children's Hospital ("KKH"), the main tertiary women and children hospital in Singapore. User acceptance of Aingeal and the Surveillance System will be considered within the clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients, aged 21 years or over
* Patients admitted to post-operative gynaecological ward at KKH Women's and Children's Hospital, Singapore
* Patients receiving opioid therapy via patient controlled analgesia (PCA)
* Patients that are on electronic nursing charting
* Patients that are on acute pain service monitoring

Exclusion Criteria:

* Patients with active, implantable devices (such as a pacemaker or ICD)
* Patients with any skin condition or injury affecting the electrode placement site
* Patients that are pregnant (Heart Rate detection algorithm has not been designed to reject foetal heart rate)

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women receiving gynaecological surgery in the mentioned hospital will be recruited.
Enrollment: 39 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Respiratory alarm rate per patient per day | 3-4 days (upon admission till 1-3 days after surgery)
  De-identified log files will be extracted from the Surveillance Station and reprocessed to produce counts of the number of respiratory alarms raised during monitoring. A sample of the data will be reviewed against the nursing chart to determine whether respiratory alarms are defined as True or False, with an overall Alarm Rate per patient per day derived.

SECONDARY OUTCOMES:
Overall Cardiac alarm rate per patient per day | 3-4 days (upon admission till 1-3 days after surgery)
  De-identified log files will be extracted from the Surveillance Station and reprocessed to produce counts of the number of cardiac alarms raised during monitoring. A sample of the data will be reviewed against the nursing chart to determine whether cardiac alarms are defined as True or False, with an overall Alarm Rate per patient per day derived.
False positive Respiratory alarm rate per patient per day | 3-4 days (upon admission till 1-3 days after surgery)
  De-identified log files will be extracted from the Surveillance Station and reprocessed to produce counts of the number of respiratory alarms raised during monitoring. A sample of the data will be reviewed against the nursing chart to determine whether respiratory alarms are defined as True or False, with False Positive Alarm Rate per patient per day derived.
False positive Cardiac alarm rate per patient per day | 3-4 days (upon admission till 1-3 days after surgery)
  De-identified log files will be extracted from the Surveillance Station and reprocessed to produce counts of the number of cardiac alarms raised during monitoring. A sample of the data will be reviewed against the nursing chart to determine whether cardiac alarms are defined as True or False, with False Positive Alarm Rate per patient per day derived.

CONTACTS AND LOCATIONS:
Overall Officials: Ban Leong Sng, FANZCA, Study Director — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/18/NCT03750318/Prot_SAP_000.pdf